CLINICAL TRIAL: NCT06357507
Title: Molecular Characterization of Moraxella Catarrhalis Isolates From Pneumonic Children at Pediatric Assiut University Hospital
Brief Title: Molecular Characterization of Moraxella Catarrhalis From Pneumonic Children at Pediatric Assiut University Hospital
Acronym: Mcatarrhalis
Status: Not yet recruiting | Type: Observational
Sponsor: Assiut University (Other)
Responsible Party: Principal Investigator, Hayam Hamdy Mahmoud, faculty of medicine meical microbiology and immunology, Assiut University
Other Study IDs: hayam hamdy
Record Dates: First submitted 2024-04-05; First posted 2024-04-10 (Actual); Last update posted 2024-04-16 (Actual); Status verified 2024-04

CONDITIONS: Respiratory Tract Infections
MeSH Terms: conditions — Respiratory Tract Infections

STUDY DESIGN:
Observational Model: Case-Only | Time Perspective: Cross-Sectional
Biospecimen Retention: Samples With DNA — sputum samples for DNA extraction and PCR
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

SUMMARY:
moraxella catarrhalis is responsible for respiratory tract infection in children and adults with streptococcus pneumonia and haemophilus influenza.Moraxella catarrhalis is gram negative diplococci, non-motile and non spore bearing bacteria. Until, 1995 it was considered as a non pathogenic respiratory tract flora.This bacteria is an important pathogen and a common cause of both upper and lower respiratory tract infections, pneumonia, sinusitis and conjunctivitis in infants, children and in elderly patients. In adults, M. catarrhalis also causes chronic obstructive pulmonary disease (COPD) and pneumonia. However, it is associated with a number of respiratory infections affecting both children and adults, including laryngitis, bronchitis and pneumonia .

DETAILED DESCRIPTION:
This institution is polymicrobial community with other pathogens such as Streptococcus pneumoniae and Haemophilus influenza (Sethi and Murphy, 2008). The pathogenicity of M. catarrhalis is mediated by several virulence genes, including the ubiquitous surface protein genes A1 (uspA1) and A2 (uspA2), which encode virulence factors that promote colonization and successful host infections (Bernhard S et al.,2012).Bacterium was first isolated in 1896, it was considered to be a harmless commensal of the upper respiratory tract for a long period of time. The bacterium rapidly colonizes the nasopharynx soon after birth asymptomatically (Blakeway et al., 2017).

ELIGIBILITY:
Inclusion Criteria:

* all children with bacterial pneumonia

Exclusion Criteria:

* viral pneumonia , tuberculosis and immunocompromised

Min Age: 1 Month | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Study Population: children with respiratory tract infection
Sampling Method: Probability Sample
Enrollment: 90 (Estimated)
Dates: Start 2024-12-01 (Estimated); Primary Completion 2027-12-01 (Estimated); Study Completion 2027-12-20 (Estimated)

PRIMARY OUTCOMES:
isolation of moraxella catarrhalis | 3 years
  isolation of organism on muller hinton agar

SECONDARY OUTCOMES:
detection of virulence genes of moraxella catarrhalis | 3 years
  detection of virulence genes by PCR
detetion of antibiotic resistance | 3years
  detetion of antibiotic resistance by agar disc diffusion

IPD SHARING:
Plan to Share IPD: No
ethical consideration

REFERENCES:
- [Background] Sethi S, Murphy TF. Infection in the pathogenesis and course of chronic obstructive pulmonary disease. N Engl J Med. 2008 Nov 27;359(22):2355-65. doi: 10.1056/NEJMra0800353. No abstract available. PMID 19038881
- [Background] Blakeway LV, Tan A, Peak IRA, Seib KL. Virulence determinants of Moraxella catarrhalis: distribution and considerations for vaccine development. Microbiology (Reading). 2017 Oct;163(10):1371-1384. doi: 10.1099/mic.0.000523. Epub 2017 Sep 12. PMID 28893369
- [Background] Bernhard S, Spaniol V, Aebi C. Molecular pathogenesis of infections caused by Moraxella catarrhalis in children. Swiss Med Wkly. 2012 Oct 29;142:w13694. doi: 10.4414/smw.2012.13694. eCollection 2012. PMID 23136074